CLINICAL TRIAL: NCT00102960
Title: A Phase III, Randomized, Open-Label Trial to Evaluate Strategies for Providing Antiretroviral Therapy to Infants Shortly After Primary Infection in a Resource Poor Setting
Brief Title: Anti-HIV Drugs for Treating Infants Who Acquired HIV Infection at Birth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIPRA ZA 002; 10404 (Registry Identifier: DAIDS ES); CHER (Registry Identifier: DAIDS ES); 5R01AI062512-02 (NIH); CIPRA-SA Project 2 (Other: CIPRA)
Record Dates: First submitted 2005-02-04; First posted 2005-02-07 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Infant; Perinatal; HIV; Disease Transmission, Vertical; Anti-Retroviral Agents; Treatment Interruption; Treatment Naive; Acute Infection; Mother-to-Child Transmission
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Didanosine; efavirenz; Lamivudine; Lopinavir; lopinavir-ritonavir drug combination; Nevirapine; Zidovudine

STUDY DESIGN:
Intervention Model Description: This study had two parts: Part A where children were enrolled with CD4% ≥ 25% and Part B where children were enrolled with CD4% < 25%. Part A had three arms: ART-Deferred, ART-40W and ART-96W where ART-40W and ART-96W were the early therapy arms for 40 and 96 weeks respectively. Part B were enrolled into two Arms: ART-40W and ART-96W. The primary efficacy analysis for CHER was based on 377 children that were enrolled in Part A in the first phase of the study. The NIH African data safety and monitoring board recommended that primary analysis be focussed on 377 children enrolled in the first phase of Part A. Additionally, all the key manuscripts have been analysed using this group. Hence all the results presented in clinicaltrials.gov will be specific to this group with three arms.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Deferred therapy Arm (Experimental): Zidovudine: First Line Regimen: Given twice daily at a dose of 240 mg/m^2 of body surface area. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2 Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line, once daily Nevirapine: Second Line, once daily
  Interventions: Drug: Abacavir sulfate; Drug: Didanosine; Drug: Efavirenz; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nevirapine; Drug: Zidovudine
- Early therapy for 40 weeks (Experimental): Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line, once daily Nevirapine: Second Line, once daily
  Interventions: Drug: Abacavir sulfate; Drug: Didanosine; Drug: Efavirenz; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nevirapine; Drug: Zidovudine
- Early therapy for 96 weeks (Experimental): Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2 Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line, once daily Nevirapine: Second Line, once daily
  Interventions: Drug: Abacavir sulfate; Drug: Didanosine; Drug: Efavirenz; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nevirapine; Drug: Zidovudine

INTERVENTIONS:
Drug: Abacavir sulfate — Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Other Names: ABC; Ziagen
Drug: Didanosine — Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age. Guidelines for switching from first line to second line therapy are available in the protocol.
  Other Names: ddI; Videx
Drug: Efavirenz — Second Line Regimen: taken orally once daily. Dosage depends on weight. Guidelines for switching from first line to second line therapy are available in the protocol.
  Other Names: EFV; Stocrin
Drug: Lamivudine — First Line Regimen: 4 mg/kg taken orally twice daily
  Other Names: 3TC; Epivir
Drug: Lopinavir/Ritonavir — First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Other Names: LPV/r; Kaletra
Drug: Nevirapine — Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Other Names: NVP; Viramune
Drug: Zidovudine — First Line Regimen: 240 mg/m^2 taken orally twice daily
  Other Names: AZT; Retrovir

SUMMARY:
The purpose of this study is to compare the effects of anti-HIV drug courses of different lengths in infants who became HIV infected at birth.

DETAILED DESCRIPTION:
In South Africa, an estimated 250,000 infants are born to HIV-infected mothers each year. A high percentage of perinatal HIV infections are due to inadequate or absent mother-to-child transmission prophylaxis. Unfortunately, even with optimal prophylaxis, relatively large numbers of HIV-infected infants will continue to be born and will require antiretroviral therapy (ART). Determining the appropriate times for initiating and interrupting treatment to benefit long-term prognosis in infants is a significant health challenge. Evidence suggests that starting ART early during acute infection will provide long-term benefits. However, longer duration of treatment increases the chance of developing drug-resistant virus, and continuous therapy begun early leads to long-term complications in children. This study will evaluate the efficacy of two different short-course ART strategies in HIV-infected infants from South Africa.

This study will last at least 3.5 years. There are two parts to this study. In Part A, infants with a baseline CD4 percentage (CD4%) of at least 25% and HIV infection diagnosed between 6 and 12 weeks of age will be randomly assigned to one of two treatment strategy arms. Arm 2 infants will receive ART for approximately 40 weeks until their first birthday. Arm 3 infants will receive ART for approximately 96 weeks until their second birthday. Treatment in both arms of Part A will begin with first-line, continuous treatment of zidovudine, lamivudine, and lopinavir/ritonavir. Those who were initially deferred treatment in Arm 1 will be reassessed for initiation of first-line, continuous ART.

First-line ART will be started in Arm 1 or restarted after interruption in Arms 2 and 3 if the appropriate criteria as defined in the protocol is met. First-line treatment of zidovudine, lamivudine, and lopinavir/ritonavir will continue until infants reach a study endpoint; when this occurs, infants will then change to second-line therapy. Second-line ART will consist of didanosine, abacavir sulfate, nevirapine and efavirenz.

All the primary efficacy analysis for this study will focus on the children enrolled in the first phase of Part A (n=377) as proposed by the data safety and monitoring board.

Follow-up visits will take place for 3.5 to 5 years, depending on time of enrollment. All infants will receive routine immunizations and cotrimoxazole (sulfamethoxazole/trimethoprim) prophylaxis from age 6 weeks until Week 40. Study visits will occur at study entry, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48; and every 12 weeks thereafter. At these visits, infants will have vital sign measurements, a physical exam, and a medical history evaluation. Blood and urine collection will occur at all study visits. Infants' parents or guardians will also be asked to complete an adherence questionnaire.

Participants enrolled in CIPRA-ZA Project 2 are encouraged to enroll in an observational substudy organized by the Wistar Institute (Dr. Luis Montaner, Principal Investigator), in conjunction with the CIPRA team. This study is entitled,"Pediatric Immune Correlates of Early Anti-HIV Therapy." The goal of this 5-year substudy is to evaluate 120 HIV infected children from the parent study twice a year and compare them to HIV uninfected age-matched controls. Children will be evaluated by (a) characterization and identification of the innate and adaptive immune reconstitution outcomes of early (9 or 21 months) therapy in infants infected with HIV at birth and (b) identification of immune correlate outcomes to clinical progression within a period of 2 to 3 years of follow-up after stopping therapy.

ELIGIBILITY:
Inclusion Criteria for Infants:

NOTE: Per Letter of Amendment dated 04/04/07, Part B of this study is no longer recruiting participants. Per Letter of Amendment dated 09/16/08 Arm 1 of this study is longer recruiting.

* HIV infected
* Antiretroviral naive. Infants who have previously received antiretroviral drugs used to prevent mother-to-child transmission are eligible for the study.
* Parent or legal guardian willing to provide informed consent and comply with study requirements

Exclusion Criteria for Infants:

* Any major life-threatening congenital abnormalities
* Severe CDC Stage B or C disease
* Liver enzyme, absolute neutrophil count, hemoglobin, electrolyte, creatinine, or clinical toxicity of Grade 3 or higher at screening
* Any acute or clinically significant medical event that would preclude participation in the study. Randomization can take place as soon as the incurrent illness has resolved if the child is still less than or equal to 12 weeks of age.
* Use of investigational drugs
* Require certain medications. More information on this criterion can be found in the protocol.
* Inability to tolerate oral medication
* Birth weight less than 2 kg (4.4 lbs)

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 377 (Actual)
Dates: Start 2005-07; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McIntyre, MBChB, MRCOG, Principal Investigator — Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, University of the Witwatersrand; Avy Violari, MBChB, FCPSA, Study Chair — Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, University of the Witwatersrand; Mark F. Cotton, PhD, Study Chair — Department of Pediatrics and Child Health, Faculty of Health Sciences, University of Stellenbosch

IPD SHARING:
Plan to Share IPD: No
Data may be made available through a formal request to the protocol team

REFERENCES:
- [Background] Faye A, Bertone C, Teglas JP, Chaix ML, Douard D, Firtion G, Thuret I, Dollfus C, Monpoux F, Floch C, Nicolas J, Vilmer E, Rouzioux C, Mayaux MJ, Blanche S; French Perinatal Study. Early multitherapy including a protease inhibitor for human immunodeficiency virus type 1-infected infants. Pediatr Infect Dis J. 2002 Jun;21(6):518-25. doi: 10.1097/00006454-200206000-00008. PMID 12182375
- [Background] Faye A, Le Chenadec J, Dollfus C, Thuret I, Douard D, Firtion G, Lachassinne E, Levine M, Nicolas J, Monpoux F, Tricoire J, Rouzioux C, Tardieu M, Mayaux MJ, Blanche S; French Perinatal Study Group. Early versus deferred antiretroviral multidrug therapy in infants infected with HIV type 1. Clin Infect Dis. 2004 Dec 1;39(11):1692-8. doi: 10.1086/425739. Epub 2004 Nov 5. PMID 15578372
- [Background] Havens PL, Waters D. Management of the infant born to a mother with HIV infection. Pediatr Clin North Am. 2004 Aug;51(4):909-37, viii. doi: 10.1016/j.pcl.2004.03.004. PMID 15275981
- [Background] King SM; American Academy of Pediatrics Committee on Pediatric AIDS; American Academy of Pediatrics Infectious Diseases and Immunization Committee. Evaluation and treatment of the human immunodeficiency virus-1--exposed infant. Pediatrics. 2004 Aug;114(2):497-505. doi: 10.1542/peds.114.2.497. PMID 15286240
- [Derived] Mutsaerts EAML, Nunes MC, van Rijswijk MN, Klipstein-Grobusch K, Otwombe K, Cotton MF, Violari A, Madhi SA. Measles Immunity at 4.5 Years of Age Following Vaccination at 9 and 15-18 Months of Age Among Human Immunodeficiency Virus (HIV)-infected, HIV-exposed-uninfected, and HIV-unexposed Children. Clin Infect Dis. 2019 Aug 1;69(4):687-696. doi: 10.1093/cid/ciy964. PMID 30418528
- [Derived] Payne H, Mkhize N, Otwombe K, Lewis J, Panchia R, Callard R, Morris L, Babiker A, Violari A, Cotton MF, Klein NJ, Gibb DM. Reactivity of routine HIV antibody tests in children who initiated antiretroviral therapy in early infancy as part of the Children with HIV Early Antiretroviral Therapy (CHER) trial: a retrospective analysis. Lancet Infect Dis. 2015 Jul;15(7):803-9. doi: 10.1016/S1473-3099(15)00087-0. Epub 2015 Jun 1. PMID 26043884
- [Derived] Cotton MF, Violari A, Otwombe K, Panchia R, Dobbels E, Rabie H, Josipovic D, Liberty A, Lazarus E, Innes S, van Rensburg AJ, Pelser W, Truter H, Madhi SA, Handelsman E, Jean-Philippe P, McIntyre JA, Gibb DM, Babiker AG; CHER Study Team. Early time-limited antiretroviral therapy versus deferred therapy in South African infants infected with HIV: results from the children with HIV early antiretroviral (CHER) randomised trial. Lancet. 2013 Nov 9;382(9904):1555-63. doi: 10.1016/S0140-6736(13)61409-9. PMID 24209829
- [Derived] Hainline C, Taliep R, Sorour G, Nachman S, Rabie H, Dobbels E, van Rensburg AJ, Cornell M, Violari A, Madhi SA, Cotton MF. Early Antiretroviral Therapy reduces the incidence of otorrhea in a randomized study of early and deferred antiretroviral therapy: Evidence from the Children with HIV Early Antiretroviral Therapy (CHER) Study. BMC Res Notes. 2011 Oct 26;4:448. doi: 10.1186/1756-0500-4-448. PMID 22029910
- [Derived] Violari A, Cotton MF, Gibb DM, Babiker AG, Steyn J, Madhi SA, Jean-Philippe P, McIntyre JA; CHER Study Team. Early antiretroviral therapy and mortality among HIV-infected infants. N Engl J Med. 2008 Nov 20;359(21):2233-44. doi: 10.1056/NEJMoa0800971. PMID 19020325

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results are presented for only 377 participants that were enrolled into the three arms (ART-Def 125, ART-40W 126 and ART-96W 126).
Groups:
- ART-Deferred: For participants with a CD4% of at least 25%, ART deferred until necessary. Once ART therapy was initiated, it was taken continously.
  Zidovudine: First Line Regimen: Given twice daily at a dose of 240 mg/m^2 of body surface area. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
- Early ART up to 40 Weeks: For participants with a CD4% of at least 25%, receive 40 weeks of ART until first birthday
  Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
- Early ART up to 96 Weeks: For participants with a CD4% of at least 25%, receive ART for 96 weeks until second birthday
  Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
Period: Overall Study
Arm/Group | ART-Deferred | Early ART up to 40 Weeks | Early ART up to 96 Weeks
Started | 125 | 126 | 126
Completed | 95 | 103 | 98
Not Completed | 30 | 23 | 28
Not completed — Death | 23 | 11 | 11
Not completed — Lost to Follow-up | 6 | 12 | 16
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Deferred Therapy: For participants with a CD4% of at least 25%, ART deferred until necessary. Once ART therapy was initiated, it was taken continously.
  Zidovudine: First Line Regimen: Given twice daily at a dose of 240 mg/m^2 of body surface area. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
- Early Therapy up to 40 Weeks: For participants with a CD4% of at least 25%, receive 40 weeks of ART until first birthday
  Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
- Early Therapy up to 96 Weeks: For participants with a CD4% of at least 25%, receive ART for 96 weeks until second birthday
  Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
- Total: Total of all reporting groups
Arm/Group | Deferred Therapy | Early Therapy up to 40 Weeks | Early Therapy up to 96 Weeks | Total
Number analyzed (Participants) | 125 | 126 | 126 | 377
Age, Continuous [Median (Inter-Quartile Range); unit: Weeks] | 7.1 [6.4 to 8.9] | 7.4 [6.6 to 8.7] | 7.5 [6.6 to 9.0] | 7.3 [6.5 to 8.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 76 | 74 | 220
  Male | 55 | 50 | 52 | 157
Region of Enrollment [Number; unit: Participants]
  South Africa | 125 | 126 | 126 | 377

OUTCOME MEASURES:

1. Primary Outcome: Time to Failure of First Line Therapy or Death
Description: To compare time to failure of first line ART (due to clinical, virological or immunological disease progression, or regimen-limiting ART toxicities) or death among three randomized arms (infants who receive early ART in Arms 2 and 3 and infants in whom ART is deferred until clinical or immunological disease progression in Arm 1) during the study (up to 4.8 years). The number of participants experiencing the events did not reach the 50% survival and thus median time-to-event is not be presented. Therefore we report the number of participants experiencing the events per Arm.
Time Frame: From date of randomization up to failure of first-line therapy or death from any cause, whichever came first, assessed up to 4.8 years
Population: In the analysis of failure of first-line therapy, children enrolled in the ART-Deferred group were used as the reference category in the hazard ratio analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Deferred Therapy: For participants with a CD4% of at least 25%, ART deferred until necessary. Once ART therapy was initiated, it was taken continuously.
  Zidovudine: First Line Regimen: Given twice daily at a dose of 240 mg/m^2 of body surface area. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
Arm/Group | Deferred Therapy | Early Therapy up to 40 Weeks | Early Therapy up to 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Participants | 48 | 32 | 26
Statistical Analysis 1: Comparison: Deferred Therapy vs Early Therapy up to 40 Weeks; Statistical analysis compares early therapy 40 weeks (ART-40W) relative to deferred therapy (ART-Def); Test type: Superiority or Other; p = 0.02, Regression, Cox; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.38 to 0.93]
Statistical Analysis 2: Comparison: Deferred Therapy vs Early Therapy up to 96 Weeks; Statistical analysis compares early therapy 96 weeks (ART-96W) relative to deferred therapy (ART-Def); Test type: Superiority or Other; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.27 to 0.76]

2. Primary Outcome: Number of Participants Who Experienced Immunological Failure Defined as Failure of CD4% to Reach 20% or CD4% Falls Below 20% on Two Occasions, Within 4 Weeks, at Any Time After the First 24 Weeks of Therapy (Initial Therapy or Restart)
Description: This was part of the primary outcome measure above. The primary outcome was a composite endpoint. The primary outcome analysis only considered the initially enrolled children that were 377 in total (ART-Deferred n=125, Early therapy 40 weeks n=126 and Early therapy 96 weeks n=126). This was part of the primary outcome measure that was a composite endpoint.
Time Frame: This outcome was assessed from the date of randomization to immunological failure. Immunological failure was assessed in the entire study duration of 4.8 years.
Measure: Count of Participants; unit: Participants
Groups:
- Early ART for 40 Weeks: For participants with a CD4% of at least 25%, receive 40 weeks of ART until first birthday
  Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
- Early Therapy for 96 Weeks: For participants with a CD4% of at least 25%, receive ART for 96 weeks until second birthday
  Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily
Arm/Group | Deferred Therapy | Early ART for 40 Weeks | Early Therapy for 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Participants | 9 | 14 | 11

3. Primary Outcome: Number of Participants Who Experienced Regimen-limiting ART Drug Toxicity
Description: Development of toxicity requiring more than one drug substitution within the same class or a switch to a new class of drugs (regimen-limiting toxicity failure) or requiring a permanent treatment discontinuation. This was part of the primary outcome measure that was a composite endpoint.
Time Frame: Regimen limiting drug toxicity was monitored from randomization up to the entire study duration of 4.8 years.
Measure: Count of Participants; unit: Participants
Groups:
- Early Therapy 40 Weeks: For participants with a CD4% of at least 25%, receive 40 weeks of ART until first birthday
  Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
- Early Therapy 96 Weeks: For participants with a CD4% of at least 25%, receive ART for 96 weeks until second birthday
  Zidovudine: First Line Regimen: 10 mg/mL taken orally twice per day. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Experienced Clinical Failure (Defined as Development of Severe CDC Stage B or Stage C Disease.) on Therapy.
Description: This included development of severe CDC Stage B or Stage C disease.This was part of the primary outcome measure that was a composite endpoint
Time Frame: Clinical failure on therapy was assessed at each visit for the entire study duration of 4.8 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Participants | 8 | 6 | 5

5. Primary Outcome: Number of Participants Who Experienced Virological Failure Defined as Confirmed HIV-1 RNA Value of at Least 10,000 Copies Per/ml Recorded on Two Consecutive Separate Occasions After 24 Weeks of Treatment (Initial Therapy or Restart)
Description: This was part of the primary outcome measure that was a composite endpoint that included confirmed HIV-1 RNA value of at least 10,000 copies per/ml recorded on two consecutive separate occasions after 24 weeks of treatment (initial therapy or restart).
Time Frame: Virological failure was assessed from randomization through the entire study duration of 4.8 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Participants | 10 | 1 | 1

6. Secondary Outcome: Number of Children Experiencing Severe CDC Stage B or Stage C Disease or Death (Cumulative After 3.5 Years)
Description: The outcome measure is defined as a number because it represents the number of children that experienced severe CDC Stage B or Stage C disease or death as defined in the outcome measure title above
Time Frame: Occurrence of severe CDC Stage B or Stage C disease or death (cumulative after 3.5 years), whichever came first, was assessed from randomization up to at least 3.5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Participants | 41 | 28 | 21
Statistical Analysis 1: Comparison: Deferred Therapy vs Early Therapy 40 Weeks; Relative to ART-Def, ART-40W had a 13% difference in the cumulative probability of clinical disease progression or death at 3·5 years; Test type: Superiority or Other; p = 0.03, Proportion test; Kaplan-Meier Cummulative Probability = 0.13, 95% CI 2-sided [0.01 to 0.25]
Statistical Analysis 2: Comparison: Deferred Therapy vs Early Therapy 96 Weeks; Relative to ART-Def, ART-96W had a 13% difference in the cumulative probability of clinical disease progression or death at 3·5 years; Test type: Superiority; p = 0.0006, Proportion test; Kaplan-Meier Cummulative Probability = 0.20, 95% CI 2-sided [0.09 to 0.31]

7. Secondary Outcome: Total Occurrence of Grade 3 or 4 Clinical Events
Description: This was a secondary outcome measure that assessed the total count of Grade 3 or 4 (clinical or laboratory) adverse events.
Time Frame: 4.8 years
Population: This analysis was only performed on the primary groups including a total of 377 participants
Measure: Number; unit: Count of events
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Count of events | 170 | 118 | 88
Statistical Analysis 1: Comparison: Deferred Therapy vs Early Therapy 40 Weeks vs Early Therapy 96 Weeks; The CHER study compared Grade 3 or 4 clinical event rates per 100 person-years between the three arms using Poisson regression modeling over the study duration of 4.8 years; Test type: Superiority or Other; p < 0.0001, Poisson Regression — This p-value compares event rates per 100 person-years across the three arms; Rate per 100 person years = 0; The rates per 100 person-years were 33.8 (Arm 1), 21.6 (Arm 2) and 16 (Arm 3)

8. Secondary Outcome: Total Occurrence of Grade 3 or 4 Laboratory Events
Time Frame: From randomization up to 4.8 years
Measure: Number; unit: Count of events
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Count of events | 35 | 44 | 33
Statistical Analysis 1: Comparison: Deferred Therapy vs Early Therapy 40 Weeks vs Early Therapy 96 Weeks; The event rates per 100 person years were compared across the three arms; Test type: Superiority; p = 0.46, Poisson regression; Rate per 100 person years = 0; The laboratory events per 100 person years across the three arms were: 7 (Deferred arm), 8.1 (early therapy for 40 weeks) and 6 (early therapy for 96 weeks)

9. Secondary Outcome: Time From Randomization to Starting or Needing to Start Continuous Therapy
Description: Time from randomization to starting (deferred therapy Arm) or needing to start continuous therapy (early therapy 40 or 96 weeks)
Time Frame: 4.8 years
Measure: Median (Full Range); unit: Weeks
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Weeks | 20 [16 to 25] | 33 [26 to 45] | 70 [35 to 109]

10. Secondary Outcome: Number of Participants With Indicated Viral Resistance Mutations at the Time of Failure of First Line Therapy
Description: Resistance testing was performed on samples with a VL≥1000 c/ml together with the matched baseline sample, if available. Reverse transcriptase (NRTI and NNRTI) and protease (PI) inhibitor mutations were analysed using a validated in-house population-based sequencing assay and the IAS 2011 mutation list.
Time Frame: 4.8 years
Population: Mutations presented descriptively were 1) Protease inhibitor mutations and 2) Met184Val mutations were reported. Only 32 participants with viral load above 1,000 copies/ml at their last visit while on treatment were analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 5 | 14 | 13
Participants
  PI mutations | 1 | 1 | 0
  Met184Val mutations | 1 | 5 | 1
  No mutations | 3 | 8 | 12

11. Secondary Outcome: Time to Death Alone or Death Plus Life Threatening Stage C Events or HIV Events Associated With Permanent End-organ Damage.
Description: This was a composite endpoint in which the number of children experiencing the events is reported. The number of participants experiencing the events did not reach the 50% survival and thus median time-to-event is not be presented. Therefore, we report the number of participants experiencing the events per Arm.
Time Frame: 4.8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Participants | 34 | 18 | 13
Statistical Analysis 1: Comparison: Deferred Therapy vs Early Therapy 40 Weeks; The analysis compares ART-40W relative to the ART-Def arm; Test type: Superiority or Other; p = 0.011, Regression, Cox; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.27 to 0.84] — Hazard rate reported above compares early therapy 40 weeks relative to the deferred therapy arm
Statistical Analysis 2: Comparison: Deferred Therapy vs Early Therapy 96 Weeks; The analysis compares ART-96 Weeks relative to ART-Deferred; Test type: Superiority or Other; p = 0.0009, Regression, Cox; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.18 to 0.64] — The hazard ratio compares ART-96W relative to the ART-Def arm

12. Secondary Outcome: Hospitalization Rates
Description: Hospitalisation rates in the three arms enrolled in the CHER study
Time Frame: 4.8 years
Measure: Number; unit: Events per 100 person years
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Events per 100 person years | 27.6 | 16.4 | 14.2

13. Secondary Outcome: Duration of Hospitalisation
Description: This is the total number of days spent in hospital by the participants and is reported per arm
Time Frame: 4.8 years, the study duration
Measure: Number; unit: Days
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Days | 1018 | 533 | 414
Statistical Analysis 1: Comparison: Deferred Therapy vs Early Therapy 40 Weeks vs Early Therapy 96 Weeks; Test type: Superiority; p = 0.004, Poisson regression — The p-value here compares the days spent in hospital across the three arms; Count of days = 0; The total number of days/count of days: 1018 (Arm 1), 533 (Arm 2) and 414 (Arm 3) were compared across the three groups by Poisson regression analysis

14. Secondary Outcome: Time to First Hospitalization
Description: To compare time to first hospitalization in the three randomized arms (infants who received early ART in Arms 2 and 3 and those who received deferred ART in Arm 1). Not all participants were hospitalized and thus the upper limits could not be evaluated.
Time Frame: From randomization up to 4.8 years
Measure: Median (Full Range); unit: Weeks
Arm/Group | Deferred Therapy | Early Therapy 40 Weeks | Early Therapy 96 Weeks
Number analyzed (Participants) | 125 | 126 | 126
Weeks | 73.1 [22.6 to NA] — Upper limit of median not estimable | NA [184.4 to NA] — The median is not estimable because the survival curve did not cross the 50% survival | NA [179.0 to NA] — The median is not estimable because the survival curve did not cross the 50% survival
Statistical Analysis 1: Comparison: Deferred Therapy vs Early Therapy 40 Weeks; Test type: Superiority; p = 0.0021, Regression, Cox; Hazard Ratio (HR) = 0.562, 95% CI 2-sided [0.389 to 0.811]
Statistical Analysis 2: Comparison: Deferred Therapy vs Early Therapy 96 Weeks; Test type: Superiority; p = 0.0038, Regression, Cox; Hazard Ratio (HR) = 0.583, 95% CI 2-sided [0.405 to 0.840]

ADVERSE EVENTS:
Time Frame: 4.8 years, the study duration
Description: Only System Organ Class and Higher Level Terms are reported for 377 participants (ART-Def 125, ART-40W 126 and ART-96W 126)
Groups:
- ART-Deferred: For participants with a CD4% of at least 25%, ART deferred until necessary. Once ART therapy was initiated, it was taken continuously.
  Zidovudine: First Line Regimen: Given twice daily at a dose of 240 mg/m^2 of body surface area. Dose was adjusted by age as the children grew older.
  Lamivudine: First Line Regimen: 4 mg/kg taken orally twice daily
  Lopinavir/Ritonavir: First Line Regimen: taken orally twice daily. Dosage depends on age and weight.
  Ritonavir: First Line Regimen taken orally twice a day. Started at 250 mg/m^2
  Abacavir sulfate: Second Line Regimen: 8 mg/kg taken orally twice daily. Guidelines for switching from first line to second line therapy are available in the protocol.
  Didanosine: Second Line Regimen: Either 100 mg/m^2 or 120 mg/m^2 taken orally twice daily. Dosage depends on age.
  Efavirenz: Second Line Regimen: taken orally once daily. Dosage depends on weight.
  Nevirapine: Second Line Regimen: 150 - 200 mg/m^2 taken orally twice daily.
Arm/Group | ART-Deferred | Early ART up to 40 Weeks | Early ART up to 96 Weeks
All-Cause Mortality (participants affected / at risk) | 23/125 | 11/126 | 11/126
Serious Adverse Events (participants affected / at risk) | 79/125 | 60/126 | 53/126
Other Adverse Events (participants affected / at risk) | 123/125 | 122/126 | 125/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ART-Deferred (N=125) | Early ART up to 40 Weeks (N=126) | Early ART up to 96 Weeks (N=126)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral palsy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing loss unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 11 (12) | 5 (5) | 2 (4)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Accidental death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Apparent death (General disorders) | 2 (2) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Unknown cause of death (General disorders) | 6 (6) | 2 (2) | 5 (5)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HIV wasting syndrome (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 5 (5) | 3 (3) | 3 (5)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 6 (8) | 4 (6) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Chickenpox (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Croup (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Cytomegalovirus encephalitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Cytomegalovirus hepatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Esophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 38 (53) | 22 (29) | 27 (31)
Laryngotracheo bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 6 (7) | 2 (2) | 2 (2)
Miliary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumococcal pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumocystis carinii pneumonia (Infections and infestations) | 5 (6) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 26 (34) | 18 (25) | 17 (20)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Septicaemia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TB (Infections and infestations) | 4 (4) | 3 (3) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculous bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4) | 0 (0)
Viral meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Burns (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fracture femur (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
AST increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma GT increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Kwashiorkor (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile seizure (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Focal seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumococcal meningitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Rectovaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ART-Deferred (N=125) | Early ART up to 40 Weeks (N=126) | Early ART up to 96 Weeks (N=126)
Lymphadenopathy (Blood and lymphatic system disorders) | 38 (46) | 52 (64) | 39 (42)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 9 (10) | 14 (17)
Splenomegaly (Blood and lymphatic system disorders) | 32 (36) | 23 (28) | 10 (14)
Gastroenteritis (Gastrointestinal disorders) | 80 (160) | 85 (214) | 81 (178)
Hepatomegaly (Hepatobiliary disorders) | 53 (72) | 50 (72) | 52 (79)
AIDS encephalopathy (Infections and infestations) | 10 (10) | 15 (15) | 10 (10)
Bronchiolitis (Infections and infestations) | 58 (83) | 66 (104) | 48 (76)
Bronchopneumonia (Infections and infestations) | 9 (10) | 12 (13) | 12 (14)
Candida nappy rash (Infections and infestations) | 17 (19) | 16 (19) | 14 (18)
Candidiasis (Infections and infestations) | 29 (41) | 32 (38) | 17 (21)
Gastroenteritis (Infections and infestations) | 52 (72) | 42 (61) | 47 (64)
Impetigo (Infections and infestations) | 27 (37) | 26 (31) | 21 (24)
Molluscum Contagiosum (Infections and infestations) | 9 (10) | 10 (11) | 10 (12)
Mucocutaneous Herpes Simplex (Infections and infestations) | 8 (9) | 7 (8) | 9 (10)
Oral Candidiasis (Infections and infestations) | 60 (101) | 46 (81) | 50 (58)
Otitis Media (Infections and infestations) | 70 (140) | 81 (220) | 78 (154)
Persistent Generalised Lymphadenopathy (Infections and infestations) | 13 (14) | 17 (19) | 21 (23)
Pharyngitis (Infections and infestations) | 69 (112) | 65 (139) | 62 (118)
Pneumonia (Infections and infestations) | 49 (81) | 44 (78) | 45 (78)
Scabies (Infections and infestations) | 13 (15) | 28 (38) | 20 (25)
TB (Infections and infestations) | 23 (24) | 28 (31) | 25 (25)
Tinea (Infections and infestations) | 49 (63) | 50 (78) | 53 (81)
Tonsilitis (Infections and infestations) | 41 (72) | 49 (89) | 39 (68)
Urinary tract infection (Infections and infestations) | 10 (12) | 15 (21) | 6 (7)
Varicella Zoster (Infections and infestations) | 7 (7) | 16 (16) | 5 (5)
ALT Increased (Investigations) | 11 (12) | 8 (10) | 4 (5)
Gamma GT Increased (Investigations) | 7 (7) | 4 (6) | 2 (3)
Failure to thrive (Metabolism and nutrition disorders) | 37 (41) | 31 (37) | 19 (23)
Dermatitis (Skin and subcutaneous tissue disorders) | 103 (320) | 96 (223) | 89 (206)
Nappy rash (Skin and subcutaneous tissue disorders) | 9 (10) | 19 (31) | 7 (10)

LIMITATIONS AND CAVEATS:
The CHER study did not include an early continuous therapy Arm, had not been powered to test for differences between early therapy 40 weeks vs. 96 weeks and never assessed in-utero vs. intrapartum infections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No